CLINICAL TRIAL: NCT06656039
Title: Development and Validation of a Multimodal Predictive Recurrence Score for Patients With Clear Cell Renal Cell Carcinoma: a Multicenter Cohort Study
Brief Title: A Multimodal Predictive Recurrence Score for Patients With Clear Cell Renal Cell Carcinoma
Status: Completed | Type: Observational
Sponsor: RenJi Hospital (Other)
Collaborators: The First Affiliated Hospital of Anhui Medical University (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); Second Affiliated Hospital of Soochow University (Other); Qianfoshan Hospital (Other); Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ccRCC MRPS
Record Dates: First submitted 2024-10-20; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Renal Cell Carcinoma, Clear Cell
Keywords: Renal Cell Carcinoma; Multimodal; Artificial Intelligence; Prognosis; Deep Learning; Multicentre Study
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — HE pathology sections of ccRCC postoperative tissues
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Training cohort
- Validation cohort
- Test cohort

SUMMARY:
The main goal of this observational study is to construct a predictive recurrence model for renal clear cell carcinoma through an artificial intelligence multimodal algorithm, which will improve the prognosis and survival time of ccRCC patients by helping clinicians to formulate individualised follow-up and to screen for appropriate adjuvant therapy candidates.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malignant renal tumours must have postoperative pathological confirmation of renal clear cell carcinoma with pathological TNM stage Ⅰ-Ⅲ;
* Have available preoperative imaging
* Have available post-operative pathological paraffin samples or HE-stained tissue sections
* Must agree to and be able to comply with the study's visit schedule and other requirements as specified in the protocol, including follow-up visits by telephone

Exclusion Criteria:

* The patient's tumour type cannot be determined on the basis of histopathological sections
* Simultaneous combination of primary tumours at other sites;
* No regular follow-up imaging data
* Cases in which other factors led the investigator to believe that enrolment was inappropriate
* Cases that met all the inclusion criteria of the appeal and did not meet all the exclusion criteria were selected for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pathologically confirmed postoperative patients with renal clear cell carcinoma of TNM stage I-III
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Disease free survival | "Baseline, immediately after the surgery", "Tumour recurrence or further follow-up", "Three months after surgery", "Six months after surgery", "Every year after surgery, at least follow-up 2years, up to 10 years"
  Defined as from surgery to tumor recurrence or follow-up deadline

CONTACTS AND LOCATIONS:
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to interested research partners upon reasonable request to Zhaiwei or Department of Urology, Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China.; the prerequisite for this is a data transfer agreement, approved by the legal departments of the requesting researcher and by all legal departments of the institutions that provided data for the study, and an ethics clearance.